CLINICAL TRIAL: NCT01577940
Title: Method Study of Bilateral Transversus Abdominis Plane (TAP) Block With 24 Hours Infusion. Extent of Sensory Block, Analgetic Effect and Lung Function in Healthy Volunteers
Brief Title: Method Study: Bilateral TAP Block With 24 Hours Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Pernille Lykke Petersen, Principal investigator, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-PLP-11; 2011-005118-13 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2012-04-16 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Pain
Keywords: Transversus abdominis plane block; postoperative pain; Postoperative pain management
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion of local anesthetic (Experimental): TAP block with 20 ml of ropivacaine 0,5%, catheter with infusion of ropivacaine 0,2% 5 ml/h 24 hours.
  Interventions: Procedure: Infusion of ropivacaine
- Infusion of saline (Placebo Comparator): TAP block with 20 ml of ropivacaine 0,5%, catheter with infusion of saline 5 ml/h 24 hours.
  Interventions: Procedure: Infusion of saline

INTERVENTIONS:
Procedure: Infusion of ropivacaine — TAP block with ropivacaine 20 ml 0,5%. Catheter with infusion of ropivacaine 0,2% 5 ml/h 24 hours on one side of the abdomen.
  Arms: Infusion of local anesthetic
Procedure: Infusion of saline — TAP block with ropivacaine 0,5% 20 ml. Catheter with infusion of saline 5 ml/h 24 hours.
  Arms: Infusion of saline

SUMMARY:
The purpose of this method study in healthy volunteers is to determine the extent of sensory block following Transversus Abdominis Plane (TAP) block with 24 hours infusion of ropivacaine versus infusion of saline. Furthermore, to determined the analgesic effect of the TAP block and the influence on the lung function.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 30 years
* written consent
* ASA 1
* BMI between 18 and 25
* males

Exclusion Criteria:

* unable to communicate in Danish
* relevant drug allergy
* alcohol or/and drug abuse
* daily intake of prescription pain medication the last 4 weeks
* pain medication in the last 48 hours
* previously operated abdominal

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in extend of sensory block from baseline (pre block) to 24 hours post block, based on 6 measurements | -15 min., 1, 4, 8, 12 and 24 hours following TAP block
  Extent of sensory block using pinprick and ice

SECONDARY OUTCOMES:
Heat pain detection threshold (abdomen) | -15 min., 1, 4, 8, 12 and 24 hours following TAP block
  Gradually heating of the skin from 32 to 52 degrees Celcius. The participant indicates the temperature where the stimulus is painful.
Heat pain detection threshold (dominant forearm) | -15 min., 1, 4, 8, 12 and 24 hours following TAP block
  Gradually heating of the skin from 32 to 52 degrees Celcius. The participant indicates the temperature where the stimulus is painful.
Long Thermal stimulation (abdomen) | -15 min., 1, 4, 8, 12 and 24 hours following TAP block
  Heating of the skin, 45 degrees Celsius 1 minute. The participant indicates pain scores on a Visuel Analog Scale from 0 (no pain) to 100 (worst imaginable)
Lung function | -15 min., 1, 4, 8, 12 and 24 hours following TAP block
  Inspiratory and expiratory force

CONTACTS AND LOCATIONS:
Overall Officials: Pernille L Petersen, MD, Principal Investigator — HOC, anesthesiology, Rigshospitalet, Copenhagen
Locations (2):
- Denmark (2):
  - HOC, anesthesiology, Rigshospitalet, Copenhagen
  - HovedOrtoCentret, Rigshospitalet, Copenhagen

REFERENCES:
- [Derived] Petersen PL, Hilsted KL, Dahl JB, Mathiesen O. Bilateral transversus abdominis plane (TAP) block with 24 hours ropivacaine infusion via TAP catheters: A randomized trial in healthy volunteers. BMC Anesthesiol. 2013 Oct 10;13(1):30. doi: 10.1186/1471-2253-13-30. PMID 24106815